CLINICAL TRIAL: NCT07265401
Title: The Effect of Salutogenic Model-Based Care on Mothers of Children Suffering From Febrile Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayça Demir Yıldırım, PhD, Associate Professor, Lecturer, Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ü.Ü. Ebe Aslıhan BAŞ
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Mothers
Keywords: Salutogenic model; Fever; Care; Fever-Related Diseases
MeSH Terms: conditions — Fever

STUDY DESIGN:
Intervention Model Description: This research was designed as an experimental study with pre-test-post-test comparisons and control groups, in order to examine the effects of Salutogenic model-based care on the individual integrity and coping strategies of mothers with febrile children.
Who Masked: Participant
Masking Description: This research was designed as an experimental study with pre-test-post-test comparisons and control groups, in order to examine the effects of Salutogenic model-based care on the individual integrity and coping strategies of mothers with febrile children.
  A total of three data collection forms were used in the research: the Personal Introduction Form, the Sense of Individual Integrity Scale, and the Coping Attitudes Assessment Scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): While applying the salutogenic care model to the mothers in the experimental group (n=45), a total of three data collection forms were used: the Personal Introduction Form, the Sense of Individual Integrity Scale, and the Coping Attitudes Assessment Scale.
  Interventions: Other: Salutogenic Care Model Training Program
- Control Group (No Intervention): While routine midwifery care was given to mothers in the control group (n=45) in the service, a total of three data collection forms were used: a Personal Introduction Form, the Sense of Individual Integrity Scale, and the Coping Attitudes Assessment Scale.

INTERVENTIONS:
Other: Salutogenic Care Model Training Program — Salutogenic Care Model Training Program This is a training program that involves meeting with the salutogenic care model in 3 sessions, providing both fever-related training and completing forms.
  1. st Interview: Comprehensibility phase; This includes providing the mother with information about fever, ensuring that she is informed about fever, the cause of fever and what she should do.
  2. nd Interview: Management phase; This includes ensuring that the mother knows which practices are effective in cases of fever, the amount, timing and frequency of medication administration, and the complications that may develop if the fever is not treated correctly.
  3. rd Interview: Meaningfulness phase; This includes ensuring that the mother does not panic during a fever, preventing her fears, and reducing her anxiety because she knows how to approach a feverish child.
  Arms: Experimental Group

SUMMARY:
This study was designed as an experimental study with pre-test-post-test comparisons and control groups, in order to investigate the effects of salutogenic model-based care on the individual integrity and coping attitudes of mothers with febrile children.

DETAILED DESCRIPTION:
The research was conducted with 90 mothers, 45 in the experimental group and 45 in the control group, with children aged 0-5 years who were diagnosed with fever and admitted to the pediatric emergency department of Zeynep Kâmil Women and Children's Diseases Education and Research Hospital between October 1, 2023 and May 1, 2024. A total of three data collection forms were used in the research: Personal Introduction Form, Individual Integrity Sense Scale, and Coping Attitudes Assessment Scale. While the salutogenic care model was applied to the mothers in the experimental group (n=45), the routine midwifery care applied in the department was given to the mothers in the control group (n=45).

ELIGIBILITY:
Inclusion Criteria:

* The child must have applied to the emergency room with a fever complaint
* Have at least a primary school level education

Exclusion Criteria:

* The child with a fever must be over 5 years old
* Having a psychological disorder

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — mothers with feverish children
Enrollment: 90 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
COPE-Coping Attitudes Assessment Scale | 6 months
  COPE-Coping Attitudes Assessment Scale "Ways of Coping" was developed by Folkman and Lazarus in 1980 and COPE was developed by Carver, Scheier and Weintraub in 1989 (Folkman et al. 1980, Wegner et al. 1987). Coping Attitudes Assessment Scale is a self-report scale consisting of 60 questions and 15 subscales. Questions are answered with the options "I never do it" (1), "I occasionally do it" (2), "I do it moderately" (3), "I do it often" (4). Each of the subscales provides information about a different coping attitude. The higher the score a person gets from the subscales provides information about which coping attitude the person uses more.
Outcome Measure | 6 months
  The Sense of Integrity Scale The Sense of Integrity Scale used in the study was developed by Antonovsky (1987) to measure the abilities of individuals to maintain their health despite stress. The first version of the SOC consists of 29 items on a 7-point Likert-type scale. Eleven items on this scale relate to "understandability," eight items to "meaningfulness," and ten items to "manageability" (Geyer 1997).
  In 1987, Antonovsky revised the existing SOC scale and developed a shorter version consisting of 13 items. In this short version, five items measure understandability, four items to "meaningfulness," and the remaining four items to "manageability," all on a 7-point Likert-type scale. The scale is a self-report scale consisting of 13 items ranging from 1 to 7. It varies between 13 and 91 points.

CONTACTS AND LOCATIONS:
Overall Officials: Ayça Demir Yıldırım, PhD, Study Director — Üsküdar University
Locations (1):
- Uskudar University, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
A research article is planned to make the individual participant data (IPD) available to other researchers.